CLINICAL TRIAL: NCT03285074
Title: The Impact of Misclassification of Obesity by Body Mass Index on Mortality in Patients With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Szu-Chun Hung, MD, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Other Study IDs: 99-IRB-016-XD
Record Dates: First submitted 2017-09-14; First posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Chronic Kidney Diseases; Obesity
Keywords: Diagnostic discordance of obesity; all-cause mortality
MeSH Terms: conditions — Renal Insufficiency, Chronic; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Unlike the general population, a higher body mass index (BMI) is associated with greater survival among patients with chronic kidney disease (CKD). However, obesity is defined as excess body fat that associated with clearly elevated health risks according to the World Health Organization. In addition, muscle wasting is prevalent among CKD subjects. Thus, we hypothesized that different definition of obesity, based on BMI or body fat percentage, might have different impact on clinical outcomes among CKD population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with non-dialysis CKD defined as estimated glomerular filtration rate (eGFR) <60 ml/min/1.73 m2

Exclusion Criteria:

* subjects with liver cirrhosis
* subjects with malignancy
* subjects with an acute cardiovascular event within the 3 months before screening for inclusion
* amputee
* pregnancy
* subjects with pacemaker
* subjects with metallic implant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with nondialysis CKD with eGFR < 60ml/min/1.73m2
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2012-12-01 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | medium follow up 4.9 years
  all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Chun Hung, MD, Principal Investigator — Division of nephrology, Taipei Tzu Chi Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sharma D, Hawkins M, Abramowitz MK. Association of sarcopenia with eGFR and misclassification of obesity in adults with CKD in the United States. Clin J Am Soc Nephrol. 2014 Dec 5;9(12):2079-88. doi: 10.2215/CJN.02140214. Epub 2014 Nov 12. PMID 25392147
- [Result] Agarwal R, Bills JE, Light RP. Diagnosing obesity by body mass index in chronic kidney disease: an explanation for the "obesity paradox?". Hypertension. 2010 Nov;56(5):893-900. doi: 10.1161/HYPERTENSIONAHA.110.160747. Epub 2010 Sep 27. PMID 20876448
- [Result] Gracia-Iguacel C, Qureshi AR, Avesani CM, Heimburger O, Huang X, Lindholm B, Barany P, Ortiz A, Stenvinkel P, Carrero JJ. Subclinical versus overt obesity in dialysis patients: more than meets the eye. Nephrol Dial Transplant. 2013 Nov;28 Suppl 4:iv175-81. doi: 10.1093/ndt/gft024. PMID 24179011
- [Derived] Lin TY, Liu JS, Hung SC. Obesity and risk of end-stage renal disease in patients with chronic kidney disease: a cohort study. Am J Clin Nutr. 2018 Nov 1;108(5):1145-1153. doi: 10.1093/ajcn/nqy200. PMID 30321257
- [Derived] Lin TY, Lim PS, Hung SC. Normal-weight obesity and clinical outcomes in nondiabetic chronic kidney disease patients: a cohort study. Am J Clin Nutr. 2018 Apr 1;107(4):664-672. doi: 10.1093/ajcn/nqy006. PMID 29635500